CLINICAL TRIAL: NCT03161496
Title: Impact of Biomarkers on Pharmacokinetics and Pharmacodynamics of Direct Oral Anticoagulants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cui Yimin (Other)
Responsible Party: Sponsor-Investigator, Cui Yimin, Director of pharmacy，M.D & Ph.D, Peking University First Hospital
Organization: Peking University First Hospital (Other)
Other Study IDs: 2016[1236]
Record Dates: First submitted 2017-05-09; First posted 2017-05-19 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Novel Oral Anticoagulants; NOACs; Rivaroxaban; Apixaban; Dabigatran; Pharmacokinetics; Pharmacodynamics; Pharmacogenomics; Accurate Medication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wild genotype: Through next generation sequencing, distinguish wild genotype of NOACs
  Interventions: Genetic: detection of genotype
- mutant genotype: Through next generation sequencing, distinguish mutant genotype of NOACs
  Interventions: Genetic: detection of genotype

INTERVENTIONS:
Genetic: detection of genotype — detection of genotype by next generation sequencing

SUMMARY:
It is general that there are many factors for individual differences of drugs in clinical application, of which genetic factors accounted for more than 20%. Novel oral anticoagulants-NOACs (include rivaroxaban, apixaban, dabigatran and so on) have advantages of convenient use and no need of monitoring, compared with the traditional vitamin K antagonist. With lack of predicted biomarkers, especially the research data of Chinese, it has the important significance in studying individual differences of NOACs in the anticoagulant efficacy and safety, through the pharmacogenomics research.

The aim of this study is to determine the polymorphism of drug metabolizing enzymes, drug transporters and drug target genes in Chinese population. By detecting the gene polymorphism, we intend to study the pharmacokinetic/ pharmacodynamics/ pharmacogenomics (PK-PD-PG) correlation of NOACs and provide scientific basis for accurate medication guide for people to use NOACs.

ELIGIBILITY:
Inclusion Criteria:

(I)Chinese Healthy Volunteers

* In accordance with the inclusion criteria for each bioequivalence trial of NOACs;
* Sign informed consent of the research;
* Complete to collect indexes of pharmacodynamics and pharmacogenomics in the cycle with control drug.

(II)Chinese Patients

* In accordance with anticoagulation indications of NOACs, include prevention of thrombosis in non valvular atrial fibrillation, prevention and treatment of deep vein thrombosis / pulmonary embolism and prevention of thrombosis after knee / hip replacement;
* More than 18 years of age, male or female;
* Never received NOACs in a month and intend to take NOACs or have received NOACs for more than one week continuously;
* sign informed consent.

Exclusion Criteria:

(I)Chinese Healthy Volunteers

* In accordance with the exclusion criteria for each bioequivalence trial of NOACs;

(II)Chinese Patients

* With history of immunodeficiency disease, including positive HIV index;
* Positive Hepatitis B surface antigen (HBsAg) and HCV index;
* Combined therapy of CYP3A4 strong inhibitors and P-gp inhibitors (e.g., systemic pyrrole antifungal agents such as ketoconazole, itraconazole, voriconazole and posaconazole; human immunodeficiency virus (HIV) - protease inhibitors such as ritonavir), CYP3A4 strong inducers and P-gp inducers (e.g., rifampicin, phenytoin, phenobarbital, carbamazepine, St. John's Wort, etc.) in 14 days before treatment with NOACs;
* Severe liver dysfunction and abnormal renal function;
* Include contraindications of NOACs, such as hypersensitivity, active bleeding, moderate or severe liver disease, previous history of intracranial hemorrhage, gastrointestinal hemorrhage in the past 6 months and major operation within 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (I)Chinese Healthy Volunteers：In accordance with the criteria of each bioequivalence trial of NOACs；150-200 cases for each drug (II)Chinese Patients：In accordance with anticoagulation indications of NOACs，never received NOACs in a month and intend to take NOACs or have received NOACs for more than one week continuously；200 cases for each drug
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of stroke or systemic embolic events (including TIA) | At 1 year
  During the observation time, record the incidence of stroke or systemic embolic events (including TIA) after NOACs(rivaroxaban, apixaban, dabigatran) administration by telephone or out-patient clinic.
Incidence of bleeding events | At 1 year
  During the observation time, record the incidence of bleeding events after NOACs(rivaroxaban, apixaban, dabigatran) administration by telephone and out-patient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.

SECONDARY OUTCOMES:
Genotype detected by next generation sequencing | pre-dose of NOACs (rivaroxaban, apixaban, dabigatran)
  Collect blood specimen before NOACs administration, then detect genotype of NOACs by next generation sequencing.
Level of anticoagulant activity assessed by anti-factor Xa activity | At baseline; at 3 hours, at 8 or 9 hours, at 12 hours for Chinese healthy volunteers, at 48 or 72 hours for Chinese patients
  Before and after rivaroxaban and apixaban administration, record anti-factor Xa activity detected by blood coagulation tests.
Level of anticoagulant activity assessed by anti-factor IIa activity | At baseline; at 2 hours, at 4 hours, at 8 hours, at 12 hours for Chinese healthy volunteers, at 72 hours for Chinese patients
  Before and after dabigatran administration, record anti-factor IIa activity detected by blood coagulation tests.
Expression level of miRNA | At baseline; at 2 or 3 hours, at 4 hours (only for dabigatran), at 8 or 9 hours, at 12 hours for Chinese healthy volunteers, at 48 or 72 hours for Chinese patients.
  Before and after NOACs administration, detect the expression level of miRNA about pharmacodynamics.
Expression level of LncRNA | At baseline; at 2 or 3 hours, at 4 hours (only for dabigatran), at 8 or 9 hours, at 12 hours for Chinese healthy volunteers, at 48 or 72 hours for Chinese patients.
  Before and after NOACs administration, detect the expression level of LncRNA about pharmacodynamics.
Incidence of stroke or systemic embolic events in the other observation times | At 1 month, 6 months and 2 years (according the actual duration of NOACs taken in patiens)
  During the other observation time, record the incidence of stroke or systemic embolic events (including TIA) after NOACs(rivaroxaban, apixaban, dabigatran) administration by telephone or out-patient clinic.
Incidence of bleeding events in the other observation times | At 1 month, 6 months and 2 years (according the actual duration of NOACs taken in patiens)
  During the other observation time, record the incidence of bleeding events after NOACs(rivaroxaban, apixaban, dabigatran) administration by telephone and out-patient clinic, including subcutaneous bleeding, gingival bleeding, gastrointestinal bleeding, intracranial hemorrhage, etc.

CONTACTS AND LOCATIONS:
Locations (17):
- China (17):
  - Anhui Provincial Hospital（The First Affiliated Hospital Of USTC）, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing HuiLongGuan Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital Of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - 900 Hospital of the Joint Logistics Team (Original name: Fuzhou General Hospital of Nanjing Militray Command), Fuzhou, Fujian
  - The 7th People's Hospital of Zhengzhou, Zhengzhou, Henan
  - The Third Hospital of Changsha, Changsha, Hunan
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - The Affiliated Hospital of Jiangnan University, or called Original Wuxi Third Hospital, Wuxi, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - the First Affiliated Hospital of Liaoning University of Traditional Chinese Medicine, Shenyang, Liaoning
  - The affiliated hospital of Inner Mongolia medical university, Hohhot, Neimenggu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Xiang Q, Wang Z, Mu G, Xie Q, Liu Z, Zhou S, Zhang H, Wang Z, Jiang J, Hu K, Zhang Y, Zhao Z, Yuan D, Guo L, Wu T, Zhang J, Wang N, Xiang J, Gu Z, Sun J, Cui Y. Genetic variants influenced the risk of bleeding and pharmacodynamics of rivaroxaban in patients with nonvalvular atrial fibrillation: A multicentre prospective cohort study. Clin Transl Med. 2023 May;13(5):e1263. doi: 10.1002/ctm2.1263. PMID 37203300
- [Derived] Zhang H, Zhang Z, Liu Z, Mu G, Xie Q, Zhou S, Wang Z, Cao Y, Tan Y, Wei X, Yuan D, Xiang Q, Cui Y. Circulating miR-320a-3p and miR-483-5p level associated with pharmacokinetic-pharmacodynamic profiles of rivaroxaban. Hum Genomics. 2022 Dec 28;16(1):72. doi: 10.1186/s40246-022-00445-5. PMID 36578040
- [Derived] Liu Z, Mu G, Xie Q, Zhang H, Jiang J, Xiang Q, Cui Y. Hemoclot Thrombin Inhibitor Assay and Expected Peak-Trough Levels of Dabigatran: A Multicenter Study. Front Cardiovasc Med. 2022 Jul 22;9:894888. doi: 10.3389/fcvm.2022.894888. eCollection 2022. PMID 35935625